CLINICAL TRIAL: NCT07039799
Title: The Effect of Virtual Reality Applications on Upper Extremity Functions in Patients With Duchenne Muscular Dystrophy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Sahra Şirvan, MSc Physiotherapist, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SSirvan
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Duchenne Muscular Dystrophy (DMD); Virtual Reality
Keywords: Duchenne Muscular Dystrophy; Virtual Reality; Upper Extremity
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality + Conventional Physiotherapy (Experimental): Participants in this group will receive a conventional physiotherapy program excluding upper extremity (UE) functional exercises. In addition, they will participate in immersive virtual reality (VR)-based rehabilitation sessions using a Meta Quest 3 headset. The VR intervention includes three custom-designed games targeting shoulder, elbow, wrist, and hand movements. These sessions will be administered twice weekly for 8 weeks, with each session lasting approximately 40 minutes. Games are tailored to each participant's functional level and designed to enhance motivation, participation, and UE motor function.
  Interventions: Behavioral: Virtual Reality + Conventional Physiotherapy
- Conventional Physiotherapy (Active Comparator): Participants in this group will receive a conventional physiotherapy program including aerobic exercises, strengthening, stretching, posture training, breathing exercises, and functional upper extremity exercises. The sessions will be delivered by physiotherapists twice per week for 8 weeks, each lasting approximately 40 minutes. No virtual reality intervention will be provided in this group.
  Interventions: Behavioral: Conventional Physiotherapy

INTERVENTIONS:
Behavioral: Virtual Reality + Conventional Physiotherapy — This intervention involves the use of fully immersive virtual reality (VR) applications delivered through the Meta Quest 3 headset, integrated with hand-tracking technology. Participants engage in three custom-designed VR games aimed at improving shoulder, elbow, wrist, and hand functions. The games are tailored to individual functional levels and include progressive difficulty. Sessions are conducted twice per week for 8 weeks, each lasting approximately 40 minutes, under the supervision of a physiotherapist. This intervention is combined with conventional physiotherapy (excluding functional upper extremity exercises).
  Arms: Virtual Reality + Conventional Physiotherapy
Behavioral: Conventional Physiotherapy — This intervention consists of a standard physiotherapy program for individuals with Duchenne Muscular Dystrophy. It includes aerobic exercises, strengthening exercises, stretching routines, postural training, respiratory exercises, and functional upper extremity exercises. The sessions are delivered by a physiotherapist twice weekly for 8 weeks, with each session lasting approximately 40 minutes.
  Arms: Conventional Physiotherapy

SUMMARY:
This study aims to evaluate the effects of fully immersive virtual reality (VR) applications on upper extremity (UE) functions in individuals diagnosed with Duchenne Muscular Dystrophy (DMD). DMD is a progressive neuromuscular disorder that leads to muscle weakness and loss of function, including the upper limbs, which are essential for daily activities and independence.

In this randomized controlled trial, 36 participants with DMD will be divided into two groups: a control group receiving conventional physiotherapy and an intervention group receiving the same physiotherapy program (excluding upper extremity exercises) combined with VR-based exercises. The VR games will be designed specifically to improve shoulder, elbow, wrist, and hand functions and will be delivered using Meta Quest 3 headsets with hand-tracking capabilities.

Both groups will receive therapy twice a week for 8 weeks. Assessments will be conducted before and after the intervention, and at follow-up, using validated tools to measure UE function, grip strength, fine motor skills, trunk control, fatigue, quality of life, and participation in daily activities.

The study aims to explore innovative rehabilitation strategies for DMD and contribute to improving the independence and quality of life of affected individuals.

DETAILED DESCRIPTION:
Duchenne Muscular Dystrophy (DMD) is a progressive genetic disorder characterized by the absence of dystrophin, leading to degeneration and weakness of skeletal muscles. While early clinical symptoms primarily affect the lower extremities, upper extremity (UE) dysfunction significantly impacts daily life and independence, especially as the disease progresses and ambulation is lost. Despite its clinical relevance, upper limb rehabilitation remains underrepresented in current treatment strategies, and there is a clear need for innovative and engaging approaches tailored to this population.

Virtual reality (VR) offers an interactive and motivating rehabilitation environment, enabling repetitive task-oriented training in a controlled and safe setting. In recent years, fully immersive VR systems have gained attention in pediatric neurorehabilitation due to their potential to improve motor function while increasing patient engagement and compliance. However, research on the application of VR in DMD, particularly targeting upper limb function, remains limited.

This study is a randomized controlled trial designed to evaluate the impact of immersive VR-based rehabilitation on UE functions in children and adolescents with DMD. A total of 36 participants will be randomly assigned to either an intervention group receiving a combination of conventional physiotherapy and VR-based upper extremity training, or a control group receiving only conventional physiotherapy including aerobic, strengthening, stretching, breathing, posture, and functional exercises.

The VR program includes three custom-developed therapeutic games targeting shoulder, elbow, wrist, and hand movements. These games will be administered using the Meta Quest 3 headset with hand-tracking technology, allowing participants to interact with the virtual environment without additional controllers. The games will be adapted to each participant's functional level, with adjustable difficulty and personalized content. Sessions will take place twice weekly for 8 weeks, with each session lasting approximately 40 minutes.

Outcome measures include standardized clinical tools to assess upper extremity performance (e.g., PUL 2.0, pinch strength, pegboard test), fine motor skills, trunk control, fatigue, health-related quality of life, and participation levels. Usability and potential side effects of VR will also be evaluated through questionnaires and observation during sessions.

The findings of this trial are expected to contribute to the evidence base supporting VR as a feasible and effective tool for enhancing upper limb function in children with DMD, and to guide future integration of digital technologies in neuromuscular rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Duchenne Muscular Dystrophy (DMD)
* Age ≥ 7 years
* Ambulatory or non-ambulatory status (both are eligible)
* Ability to follow movement instructions
* Brooke Upper Extremity Functional Rating Scale (BUEFS) level ≤ 4 (i.e., able to bring hand to mouth)

Exclusion Criteria:

* Presence of any neurological diagnosis other than DMD
* Cognitive, behavioral, or communication impairments that limit participation
* Systemic illness or condition interfering with participation
* Severe visual impairments incompatible with VR headset use
* Presence of severe contractures or deformities that prevent execution of VR-based exercises

Ages: 7 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Since Duchenne Muscular Dystrophy disease is seen in males, it was planned to include male individuals in this study.
Enrollment: 36 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Performance of the Upper Limb (PUL 2.0) Score | Baseline, 8 weeks, and 4-week follow-up
  A clinician-reported outcome measure designed to assess upper limb motor performance in individuals with Duchenne Muscular Dystrophy. It includes tasks at shoulder, mid-level, and distal levels.
Pediatric Quality of Life Inventory - Neuromuscular Module (PedsQL-NM) | Baseline, 8 weeks, and 4-week follow-up
  A participant and parent-reported instrument assessing health-related quality of life in pediatric patients with neuromuscular disorders.
Participation and Environment Measure for Children and Youth (PEM-CY) | Baseline, 8 weeks, and 4-week follow-up
  A parent-reported measure assessing children's participation and environmental support at home, school, and in the community.

SECONDARY OUTCOMES:
ABILHAND-Kids Manual Ability Scale | Baseline, 8 weeks, and 4-week follow-up
  The ABILHAND-Kids is a parent-reported questionnaire designed to measure manual ability in children with upper limb impairments. It contains 21 items scored based on perceived difficulty. Minimum score: 0; Maximum score: 42. Higher scores indicate better manual ability.
Pinch Grip Strength Using Jamar Pinch Gauge | Baseline, 8 weeks, and 4-week follow-up
  Measurement of lateral pinch strength in kilograms using a standardized hand-held dynamometer.
Nine-Hole Peg Test (9HPT) | Baseline, 8 weeks, and 4-week follow-up
  A timed performance test evaluating fine motor dexterity by measuring the time taken to place and remove pegs using each hand.
Trunk Control Measurement Scale (TCMS) | Baseline, 8 weeks, and 4-week follow-up
  The Trunk Control Measurement Scale (TCMS) is a standardized clinical tool used to assess trunk control in children with neuromotor disorders. It evaluates both static and dynamic sitting balance through 15 tasks grouped into three subscales: static sitting balance, selective movement control, and dynamic reaching.Minimum score: 0; Maximum score: 58. Higher scores indicate better trunk control.
Multidimensional Fatigue Scale (PedsQL Fatigue Scale) | Baseline, 8 weeks, and 4-week follow-up
  The Pediatric Quality of Life (PedsQL) Multidimensional Fatigue Scale is a standardized questionnaire used to assess fatigue in children and adolescents. It includes 18 items covering three subscales: General Fatigue, Sleep/Rest Fatigue, and Cognitive Fatigue. Each item is scored on a 5-point Likert scale and then linearly transformed to a 0-100 scale. Minimum score: 0; Maximum score: 100. Higher scores indicate better functioning.
Timed Upper Extremity Functional Tasks (e.g., T-shirt On/Off, Coin Pick-Up) | Baseline, 8 weeks, and 4-week follow-up
  A set of timed performance tasks evaluating the duration of functional UE activities.
System Usability Scale - Turkish Version (SUS-TR) | Post-intervention (8 weeks)
  The System Usability Scale - Turkish Version (SUS-TR) is the Turkish-adapted version of the System Usability Scale, a 10-item questionnaire used to evaluate the perceived usability of a system or product. Each item is rated on a 5-point Likert scale and converted to a composite score ranging from 0 to 100. Minimum score: 0; Maximum score: 100. Higher scores indicate better usability.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the inclusion of a pediatric and vulnerable population diagnosed with Duchenne Muscular Dystrophy (DMD). To protect participants' privacy and ensure compliance with ethical standards and data protection regulations, data sharing is not planned.

REFERENCES:
- [Background] Alemdaroglu I, Karaduman A, Yilmaz OT, Topaloglu H. Different types of upper extremity exercise training in Duchenne muscular dystrophy: effects on functional performance, strength, endurance, and ambulation. Muscle Nerve. 2015 May;51(5):697-705. doi: 10.1002/mus.24451. Epub 2015 Mar 5. PMID 25196721
- [Background] Kiper P, Federico S, Szczepanska-Gieracha J, Szary P, Wrzeciono A, Mazurek J, Luque-Moreno C, Kiper A, Spagna M, Barresi R, Cieslik B. A Systematic Review on the Application of Virtual Reality for Muscular Dystrophy Rehabilitation: Motor Learning Benefits. Life (Basel). 2024 Jun 22;14(7):790. doi: 10.3390/life14070790. PMID 39063545